CLINICAL TRIAL: NCT06093529
Title: Marker Expression in Pediatric Patients With Immune Thrombocytopenic Purpura Receiving Second Line Therapy
Brief Title: Immune Markers in Pediatric ITP on Second Line Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Mahmoud Abdelsalam, Principle Investigator, Assiut University
Other Study IDs: ITPIMMUNEMARKERS
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: ITP - Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Blood Cell Count; CD4 Lymphocyte Count

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Respondents to second-line therapy: Immune markers in ITPpatients Respondant to second line therapy
  Interventions: Diagnostic Test: complete blood count, CD3+ , CD4+ , CD8+, CD16+, CD56+, IFN-γ.
- Non-Respondents to second-line therapy: Immune markers in ITPpatients nonrespondant to second line therapy
  Interventions: Diagnostic Test: complete blood count, CD3+ , CD4+ , CD8+, CD16+, CD56+, IFN-γ.

INTERVENTIONS:
Diagnostic Test: complete blood count, CD3+ , CD4+ , CD8+, CD16+, CD56+, IFN-γ. — 1. Full history
  2. Thorough clinical examinations
  3. Laboratory investigations will include:
     1. complete blood count with focus on platelet count, platelet distribution width and mean platelet volume. Platelet count will be confirmed by direct blood film and blood smear.
     2. Measurements of CD3+, CD4+, CD8+ and natural killer cells (CD16+, CD56+) will be conducted using flow cytometry.
     3. Serum IFN-γ levels will be determined using an ELISA kit.
  4. Response to the treatment will be assessed according to The International Working Group criteria which defines Response as platelet count ≥ 30 x 10⁹/L and >2-fold increase in platelet count from baseline and absence of bleeding, measured on 2 occasions greater than 7 days apart. No response is characterized by a platelet count <30 x 10⁹/L or a less than 2-fold increase in platelet count from baseline, or the presence of bleeding.

SUMMARY:
Immune thrombocytopenia (ITP) is a common autoimmune disease characterized by low platelet count and increased risk of bleeding. It affects approximately 50 to 100 cases per million people per year, with children accounting for half of the cases.

DETAILED DESCRIPTION:
Antiplatelet factors in the plasma of ITP patients, specifically IgG, have been attributed to platelet destruction through phagocytosis or complement-mediated lysis. However, these antibodies are only present in 60-70% of ITP patients, suggesting that other mechanisms may be involved in platelet destruction.

B lymphocytes play a critical role in immune responses through antibody production, antigen presentation to T cells, and cytokine secretion. CD4+ T helper cells play a crucial role in supporting B cell development into antibody-secreting plasma cells. Furthermore, evidence of auto reactive CD4+ T cells targeting platelet epitopes has been reported.

It was found that there is clonal expansion of a particular subset of CD8+ T cells, known as terminally differentiated effector memory T cells (TEMRA cells), in refractory ITP. Furthermore, CD8+ T cells induce platelet activation and apoptosis in an antibody-independent mechanism for refractory thrombocytopenia that may be amenable to therapeutic targeting. IFN-γ is an important cytokine involved in host defence and immune regulation. It is primarily produced by T helper, cytotoxic T, and natural killer cells. Dysregulated secretion of IFN-γ has been implicated in the development of autoimmune disorders. Initial studies on ITP focused on the role of autoantibodies. Therefore, drug discovery efforts have focused on suppressing aberrant humoral immunity through B cell depletion, disruption of immunoreceptor, and inhibition of autoantibody activity. By comparing the marker expression in different treatment response groups, the investigator can potentially identify markers that may serve as predictive or prognostic indicators of treatment response. This information could be valuable for guiding treatment decisions and optimizing patient outcomes in pediatric ITP.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients diagnosed with immune thrombocytopenia who are undergoing second line therapy with either eltrombopag or romiplostim.

Exclusion Criteria:

* Include acute immune thrombocytopenic children receiving first line therapy and those with secondary immune thrombocytopenia.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with ITP who are receiving second-line therapy who are attending the outpatient pediatric hematology clinic at Assiut University Children Hospital or the clinic at Central Insurance Agency of Assiut.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Correlation analysis | One year
  Analysis of the correlation between specific markers expression ( CD3,CD4,CD8,Interferon gamma and natural killer cells) and treatment response in pediatric patients with immune thrombocytopenia who are receiving second line therapy.

SECONDARY OUTCOMES:
Assessment of treatment response | One year
  Assessment of response to second line therapy (eltrombopag, romiplostim) in pediatric patients with immune thrombocytopenic purpura using clinical and laboratory findings.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled I El-sayeh, M.D., Study Director — Assiut University; Mostafa M Embaby, M.D., Study Director — Assiut University; Azhar A Mohammed, M.D., Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kayal L, Jayachandran S, Singh K. Idiopathic thrombocytopenic purpura. Contemp Clin Dent. 2014 Jul;5(3):410-4. doi: 10.4103/0976-237X.137976. PMID 25191085
- [Background] Zufferey A, Kapur R, Semple JW. Pathogenesis and Therapeutic Mechanisms in Immune Thrombocytopenia (ITP). J Clin Med. 2017 Feb 9;6(2):16. doi: 10.3390/jcm6020016. PMID 28208757
- [Background] Cancro MP. The BLyS/BAFF family of ligands and receptors: key targets in the therapy and understanding of autoimmunity. Ann Rheum Dis. 2006 Nov;65 Suppl 3(Suppl 3):iii34-6. doi: 10.1136/ard.2006.058412. PMID 17038469
- [Background] Kuwana M, Kaburaki J, Kitasato H, Kato M, Kawai S, Kawakami Y, Ikeda Y. Immunodominant epitopes on glycoprotein IIb-IIIa recognized by autoreactive T cells in patients with immune thrombocytopenic purpura. Blood. 2001 Jul 1;98(1):130-9. doi: 10.1182/blood.v98.1.130. PMID 11418472
- [Background] Malik A, Sayed AA, Han P, Tan MMH, Watt E, Constantinescu-Bercu A, Cocker ATH, Khoder A, Saputil RC, Thorley E, Teklemichael A, Ding Y, Hart ACJ, Zhang H, Mitchell WA, Imami N, Crawley JTB, Salles-Crawley II, Bussel JB, Zehnder JL, Adams S, Zhang BM, Cooper N. The role of CD8+ T-cell clones in immune thrombocytopenia. Blood. 2023 May 18;141(20):2417-2429. doi: 10.1182/blood.2022018380. PMID 36749920
- [Background] Pollard KM, Cauvi DM, Toomey CB, Morris KV, Kono DH. Interferon-gamma and systemic autoimmunity. Discov Med. 2013 Sep;16(87):123-31. PMID 23998448
- [Background] HARRINGTON WJ, MINNICH V, HOLLINGSWORTH JW, MOORE CV. Demonstration of a thrombocytopenic factor in the blood of patients with thrombocytopenic purpura. J Lab Clin Med. 1951 Jul;38(1):1-10. No abstract available. PMID 14850832
- [Background] Shulman NR, Marder VJ, Weinrach RS. Similarities between known antiplatelet antibodies and the factor responsible for thrombocytopenia in idiopathic purpura. Physiologic, serologic and isotopic studies. Ann N Y Acad Sci. 1965 Jun 30;124(2):499-542. doi: 10.1111/j.1749-6632.1965.tb18984.x. No abstract available. PMID 5214832
- [Background] van Leeuwen EF, van der Ven JT, Engelfriet CP, von dem Borne AE. Specificity of autoantibodies in autoimmune thrombocytopenia. Blood. 1982 Jan;59(1):23-6. PMID 7032627
- [Background] Ghanima W, Khelif A, Waage A, Michel M, Tjonnfjord GE, Romdhan NB, Kahrs J, Darne B, Holme PA; RITP study group. Rituximab as second-line treatment for adult immune thrombocytopenia (the RITP trial): a multicentre, randomised, double-blind, placebo-controlled trial. Lancet. 2015 Apr 25;385(9978):1653-61. doi: 10.1016/S0140-6736(14)61495-1. Epub 2015 Feb 5. PMID 25662413
- [Background] Mahevas M, Azzaoui I, Crickx E, Canoui-Poitrine F, Gobert D, Languille L, Limal N, Guillaud C, Croisille L, Jeljeli M, Batteux F, Baloul S, Fain O, Pirenne F, Weill JC, Reynaud CA, Godeau B, Michel M. Efficacy, safety and immunological profile of combining rituximab with belimumab for adults with persistent or chronic immune thrombocytopenia: results from a prospective phase 2b trial. Haematologica. 2021 Sep 1;106(9):2449-2457. doi: 10.3324/haematol.2020.259481. PMID 32817288
- [Background] Newland AC, Sanchez-Gonzalez B, Rejto L, Egyed M, Romanyuk N, Godar M, Verschueren K, Gandini D, Ulrichts P, Beauchamp J, Dreier T, Ward ES, Michel M, Liebman HA, de Haard H, Leupin N, Kuter DJ. Phase 2 study of efgartigimod, a novel FcRn antagonist, in adult patients with primary immune thrombocytopenia. Am J Hematol. 2020 Feb;95(2):178-187. doi: 10.1002/ajh.25680. Epub 2019 Dec 10. PMID 31821591
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182